CLINICAL TRIAL: NCT04351295
Title: Clinical Study Evaluating the Efficacy of Faviprevir in COVID-19 Treatment
Brief Title: Efficacy of Faviprevir in COVID-19 Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: faviprevir covid
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: COVID
MeSH Terms: interventions — favipiravir; Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Faviprevir (Experimental): Faviprevir
  Interventions: Drug: Favipiravir
- chloroquine (Active Comparator): chloroquine
  Interventions: Drug: Chloroquine

INTERVENTIONS:
Drug: Favipiravir — Favipiravir
  Other Names: Faviprevir
  Arms: Faviprevir
Drug: Chloroquine — chloroquine oral tablets
  Arms: chloroquine

SUMMARY:
Faviprevir in COVID-19 treatment

DETAILED DESCRIPTION:
Clinical Study Evaluating the Efficacy of Faviprevir in COVID-19 treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients with covid 19

Exclusion Criteria:

* Allergy or contraindications to faviprevir

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Number of patients with mortality or need for mechanical ventilation | 6 months
  Number of patients with mortality or need for mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: sherief Abd-Elsalam, Ass. Prof., Principal Investigator — Tanta University - Faculty of Medicine
Locations (1):
- Tanta University, Ainshams University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dabbous HM, Abd-Elsalam S, El-Sayed MH, Sherief AF, Ebeid FFS, El Ghafar MSA, Soliman S, Elbahnasawy M, Badawi R, Tageldin MA. Efficacy of favipiravir in COVID-19 treatment: a multi-center randomized study. Arch Virol. 2021 Mar;166(3):949-954. doi: 10.1007/s00705-021-04956-9. Epub 2021 Jan 25. PMID 33492523 (Retraction: PMID 34811571 Arch Virol. 2022 Jan;167(1):277)